CLINICAL TRIAL: NCT00401453
Title: Carbohydrate Days as Simple and Efficient Therapy for Patients With Type 2 Diabetes Mellitus and Insulin Resistance: Oatmeal and Insulin Resistance (OMA-IR).
Brief Title: OatMeal and Insulin Resistance: OMA-IR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Alexander Lammert, Universty Hospital Mannheim
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2006-119N-MA
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Diabetes Mellitus Type 2; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

INTERVENTIONS:
Behavioral: Diet: carbohydrate days. (Name: oatmeal.) — Dietary intervention with two days of oatmeal compared to normal diabetes adapted diet in insulin resistant subjects.

SUMMARY:
Insulin resistance is a central feature of Diabetes mellitus type 2 (Stumvoll et al. 2005). Hypo- and hyperglycemic states are associated with adverse inpatient outcomes (ADA et al. 2006 Diab Care) and with the development of microvascular complications (UKPDS 34 Lancet 1998).

A long known therapy for the acute treatment of patients with deteriorated glucose metabolism and insulin resistance are carbohydrate days. The principle of the therapy was firstly introduced in 1903 by Carl von Noorden (Noorden et al. 1903). The diabetic patients were treated for several days with a carbohydrate rich diet with fat restriction. Surprisingly, this resulted in an amelioration of glucosuria. Today it's still a valuable tool for patients with uncontrollable diabetes mellitus and severe insulin resistance (Willms B. 1989). But up to now there has been no systemic evaluation of carbohydrate days in patients with deteriorated Diabetes mellitus and insulin resistance.

The investigators conducted a pilot study with 14 patients to evaluate the efficacy of two days of oatmeal on insulin resistance and glucose metabolism in an acute clinical setting and after a four week outpatient period. Inclusion criteria were type 2 diabetes with deteriorated glucose metabolism, insulin resistance defined as an insulin dosage of more than 1 U per day and kg bodyweight. Within this pilot trial the investigators found a marked decrease of insulin requirements (~40%) and mean daily blood glucose to a mean blood glucose of 114.7±36.7 mg/dl in the acute setting as well as after the four week outpatient period (Lammert et al. 2006).

The most important shortcomings of this study were the hypocaloric interventions in both groups (diabetes-adapted diet: 1500kcal/d vs. oatmeal 1200kcal/d) making it difficult to attribute the observed effects to oatmeal alone as well as the uncontrolled nature. These design flaws have been addressed within this new clinical trial. The investigators plan an open label, cross-over study with isocaloric interventions (oatmeal and diabetes-adapted diet: ~ 1200kcal/d). The intervention comprises two days of oatmeal (third and fourth day) within a 5 day hospital stay. The control is only treated with 5 days of diabetes adapted diet. Thereafter, the patients are followed every four weeks for an overall of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus 2
* insulin therapy
* stable therapy modality within the last 3 months
* deteriorated glucose metabolism (Hba1c > 7%)
* insulin resistance, defined as more than 1 unit of insulin per kg and day

Exclusion Criteria:

* acute vascular event within the last 3 months
* planed weight reducing therapy
* acute and chronic inflammatory disease
* therapy with corticosteroids
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
daily insulin requirements and glycemic control | directly before and after intervention as well as 4, 8, 12, and 16 weeks after intervention

SECONDARY OUTCOMES:
Changes in factors related to insulin resistance: | directly before and after intervention as well as 4, 8, 12, and 16 weeks after intervention
free fatty acids, leptin, sOB-R, proinsulin, uric acid, adiponectin and high molecular weight adiponectin. | directly before and after intervention as well as 4, 8, 12, and 16 weeks after intervention
Changes in markers of inflammation and macrovascular risk: | directly before and after intervention as well as 4, 8, 12, and 16 weeks after intervention
c-reactive protein, prostaglandin F2 alpha, cholesterol, HDL and LDL. | directly before and after intervention as well as 4, 8, 12, and 16 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Hammes, PhD, Study Director — fifth medical clinic, university hospital Mannheim, Theodor-Kutzer-Ufer 1-3, 68167 Mannheim, Germany; Alexander Lammert, MD, Principal Investigator — fifth medical clinic, University hospital Mannheim, Theodor-Kutzer-Ufer 1-3, 68167 Mannheim, Germany
Locations (1):
- Fifth Medical Clinic, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Stumvoll M, Goldstein BJ, van Haeften TW. Type 2 diabetes: principles of pathogenesis and therapy. Lancet. 2005 Apr 9-15;365(9467):1333-46. doi: 10.1016/S0140-6736(05)61032-X. PMID 15823385
- [Background] ACE/ADA Task Force on Inpatient Diabetes. American College of Endocrinology and American Diabetes Association Consensus statement on inpatient diabetes and glycemic control. Diabetes Care. 2006 Aug;29(8):1955-62. doi: 10.2337/dc06-9913. No abstract available. PMID 16873812
- [Background] Lammert A, Kratzsch J, Selhorst J, Humpert PM, Bierhaus A, Birck R, Kusterer K, Hammes HP. Clinical benefit of a short term dietary oatmeal intervention in patients with type 2 diabetes and severe insulin resistance: a pilot study. Exp Clin Endocrinol Diabetes. 2008 Feb;116(2):132-4. doi: 10.1055/s-2007-984456. Epub 2007 Dec 20. PMID 18095234